CLINICAL TRIAL: NCT03933748
Title: Therapeutic Drug Monitoring of Teicoplanin in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Qianfoshan Hospital (Other); Shandong Provincial Hospital (Other Government); Affiliated Hospital of Qinghai University (Other); Jinan children's hospital (Unknown); Yantai Yuhuangding Hospital (Other); Jinan Central Hospital (Other); Liaocheng People's Hospital (Other); Shandong Tumor Hospital (Other); Weifang People's Hospital (Other); Linyi People's Hospital (Other); Jining Medical University (Other); Weihai maternal and child health care hospital (Unknown); The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Other Study IDs: 2019_Teicoplanin_001
Record Dates: First submitted 2019-04-24; First posted 2019-05-01 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2019-04

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — teicoplanin-polymethylmethacrylate bead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Teicoplanin-PMMA — Therapeutic drug monitoring of teicoplanin

SUMMARY:
In this study, the therapeutic drug monitoring of teicoplanin is carried out among children to obtain the drug concentration, clinical efficacy and safety data of children patients in different gender and age groups. Then we analyze the relationship between blood drug concentration and efficacy and safety, and provide recommendations for the treatment window of teicoplanin in Chinese children.

ELIGIBILITY:
Inclusion Criteria:

* Teicoplanin was administered intravenously;
* Teicoplanin was used for therapeutic purposes;
* Age:≤18 years;
* Clinician confirms and plans to diagnose the patient with gram-positive coccus infection;
* Patients with therapeutic concentration monitoring of teicoplanin.

Exclusion Criteria:

* Teicoplanin was administered non-intravenously;
* Teicoplanin was used for prophylactic purposes;
* Patients without therapeutic concentration monitoring of teicoplanin;
* Patients who die within 24 hours of the use of teicoplanin；
* The blood concentrations of the patient was not approved by the quality control center.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with gram-positive coccus infection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentration | Through study completion, an average of 14 days
  To detect the plasma concentrations of teicoplanin at therapeutic drug monitoring (TDM).

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided